CLINICAL TRIAL: NCT01263483
Title: A Phase 2/3, Double-blind, Randomized, Placebo-controlled, Parallel-group, Multicenter Study to Determine the Efficacy and Safety of SYR-322 When Used in Combination With α-glucosidase Inhibitor in Subjects With Type 2 Diabetes in Japan
Brief Title: Efficacy and Safety of Alogliptin Used in Combination With α-glucosidase Inhibitor in Participants With Type 2 Diabetes in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322/CCT-003; U1111-1118-3955 (Registry Identifier: WHO); JapicCTI-080589 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus - Type 2; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — alogliptin; voglibose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Voglibose 0.2 mg TID (Active Comparator)
  Interventions: Drug: Voglibose
- Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID (Experimental)
  Interventions: Drug: Alogliptin and voglibose
- Alogliptin 25 mg QD and Voglibose 0.2 mg TID (Experimental)
  Interventions: Drug: Alogliptin and voglibose

INTERVENTIONS:
Drug: Alogliptin and voglibose — Alogliptin 12.5 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 12 weeks.
  Other Names: SYR-322; BASEN®; Voglibose
  Arms: Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID
Drug: Alogliptin and voglibose — Alogliptin 25 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 12 weeks.
  Other Names: SYR-322; BASEN®; Voglibose
  Arms: Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Drug: Voglibose — Alogliptin placebo-matching tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 12 weeks.
  Other Names: BASEN®
  Arms: Voglibose 0.2 mg TID

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of alogliptin, once daily (QD) combined with an α-glucosidase inhibitor taken three times daily (TID) in type 2 diabetic patients with uncontrolled blood glucose.

DETAILED DESCRIPTION:
Both insulin hyposecretion and insulin-resistance are considered to be involved in the development of type 2 diabetes mellitus.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV (DPP-IV) enzyme. DPP-IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of DPP-IV will improve glycemic control in patients with type 2 diabetes.

In Japan, α-glucosidase inhibitors are widely used as a first-line treatment for type 2 diabetes mellitus. Because alogliptin has a different mechanism of action compared to α-glucosidase inhibitors, the study evaluated the efficacy and safety of alogliptin combined with an α-glucosidase inhibitor in type 2 diabetic patients with uncontrolled blood glucose while taking a α-glucosidase inhibitor and receiving diet and/or exercise therapies.

To evaluate the long-term safety and efficacy of the concomitant use of alogliptin and an α-glucosidase inhibitor, subjects who participated in the present study could enter a long-term extension study SYR-322/OCT-003 (NCT01263509) that was planned separately.

ELIGIBILITY:
Inclusion Criteria:

* Had been receiving a stable dose and regimen of an α-glucosidase inhibitor for the last 4 weeks or longer before the start of the screening phase (Week -8) and during the screening phase.
* Had a glycosylated hemoglobin (HbA1c) value of 6.5% or more and below 10.0% 4 weeks after the start of the screening phase (Week -4).
* Had HbA1c differences within 10.0% at the start of the screening phase (Week -8) and 4 weeks after the start of the screening phase (Week -4) from the HbA1c value at the start of the screening phase.
* Was receiving a specific diet therapy and an exercise therapy (if any) for the last 4 weeks or longer before the start of the screening phase (Week -8).

Exclusion Criteria:

* Had received any antidiabetic drug other than α-glucosidase inhibitors within the last 4 weeks before the start of the screening phase (Week -8) or during the screening phase.

Ages: 33 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Department of Medicine, Study Director — Kawasaki Medical School

REFERENCES:
- [Derived] Seino Y, Fujita T, Hiroi S, Hirayama M, Kaku K. Alogliptin plus voglibose in Japanese patients with type 2 diabetes: a randomized, double-blind, placebo-controlled trial with an open-label, long-term extension. Curr Med Res Opin. 2011 Nov;27 Suppl 3:21-9. doi: 10.1185/03007995.2011.614936. PMID 22106975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at investigative sites in Japan from to .
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus with uncontrolled blood glucose despite diet and exercise therapies were enrolled in one of 3, once-daily (QD) or three-times daily (TID) treatment groups.
Groups:
- Voglibose 0.2 mg TID: Alogliptin placebo-matching tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 12 weeks.
- Alogliptin 12.5 mg QD: Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID
- Alogliptin 25 mg QD and Voglibose 0.2 mg TID: Alogliptin 25 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 12 weeks.
Period: Overall Study
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Started | 75 | 76 | 79
Completed | 68 | 74 | 74
Not Completed | 7 | 2 | 5
Not completed — Adverse Event | 4 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Participant Unavailability | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID | Total
Number analyzed (Participants) | 75 | 76 | 79 | 230
Age, Customized [Number; unit: participants]
  ≤ 64 years | 39 | 52 | 39 | 130
  ≥ 65 years | 36 | 24 | 40 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 29 | 88
  Male | 48 | 44 | 50 | 142

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Analysis based on last observation carried forward, where the last postbaseline double-blind observed value is carried forward and used for all subsequent scheduled time points where data is missing. Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 74 | 76 | 79
percentage of Glycosylated Hemoglobin | 0.04 (0.457) | -0.96 (0.553) | -0.91 (0.485)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -1.002, 95% CI 2-sided [-1.166 to -0.838]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.947, 95% CI 2-sided [-1.097 to -0.796]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 2).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 2 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 74 | 76 | 79
percentage of Glycosylated Hemoglobin | -0.01 (0.180) | -0.19 (0.149) | -0.21 (0.175)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.176, 95% CI 2-sided [-0.229 to -0.123]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.190, 95% CI 2-sided [-0.247 to -0.133]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 4).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 4 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 74 | 76 | 79
percentage of Glycosylated Hemoglobin | -0.02 (0.301) | -0.44 (0.234) | -0.43 (0.263)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.421, 95% CI 2-sided [-0.507 to -0.334]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.414, 95% CI 2-sided [-0.504 to -0.324]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 74 | 76 | 79
percentage of Glycosylated Hemoglobin | -0.01 (0.398) | -0.74 (0.427) | -0.75 (0.392)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.738, 95% CI 2-sided [-0.871 to -0.605]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.749, 95% CI 2-sided [-0.875 to -0.623]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 2).
Description: The change between the value of fasting plasma glucose collected at week 2 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 79
mg/dL | -3.5 (21.28) | -15.5 (18.77) | -18.8 (19.89)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -12.01, 95% CI 2-sided [-18.50 to -5.52]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -15.33, 95% CI 2-sided [-21.93 to -8.73]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 4).
Description: The change between the value of fasting plasma glucose collected at week 4 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 79
mg/dL | -0.6 (23.71) | -16.2 (21.84) | -22.6 (23.96)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -15.65, 95% CI 2-sided [-23.02 to -8.27]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -22.03, 95% CI 2-sided [-29.68 to -14.38]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 79
mg/dL | -2.5 (25.94) | -20.8 (22.10) | -21.9 (23.96)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -18.30, 95% CI 2-sided [-26.09 to -10.50]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -19.34, 95% CI 2-sided [-27.34 to -11.34]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 or final visit and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 79
mg/dL | -5.6 (27.87) | -19.1 (20.70) | -18.5 (25.53)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -13.53, 95% CI 2-sided [-21.46 to -5.60]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -12.97, 95% CI 2-sided [-21.53 to -4.41]

9. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 2).
Description: The change between the value of fasting C-peptide collected at week 2 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 79
ng/mL | 0.03 (0.668) | -0.07 (0.593) | -0.01 (0.599)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.100, 95% CI 2-sided [-0.304 to 0.104]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.036, 95% CI 2-sided [-0.239 to 0.167]

10. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 4).
Description: The change between the value of fasting C-peptide collected at week 4 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 79
ng/mL | 0.05 (0.753) | 0.06 (0.955) | 0.01 (0.682)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.013, 95% CI 2-sided [-0.267 to 0.292]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.034, 95% CI 2-sided [-0.264 to 0.196]

11. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 8).
Description: The change between the value of fasting C-peptide collected at week 8 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 79
ng/mL | 0.07 (0.691) | 0.03 (0.725) | -0.01 (0.468)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -0.038, 95% CI 2-sided [-0.268 to 0.191]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -0.073, 95% CI 2-sided [-0.261 to 0.115]

12. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 12).
Description: The change between the value of fasting C-peptide collected at week 12 or final visit and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 73 | 76 | 79
ng/mL | 0.02 (0.664) | 0.06 (0.680) | 0.10 (0.620)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.035, 95% CI 2-sided [-0.183 to 0.252]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [-0.124 to 0.288]

13. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value).
Description: The change between the value of blood glucose collected at week 12 or final visit and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 67 | 75 | 75
mg/dL | 72.4 (34.89) | 40.9 (23.23) | 38.7 (32.33)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -31.54, 95% CI 2-sided [-41.28 to -21.80]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -33.73, 95% CI 2-sided [-44.88 to -22.57]

14. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (AUC (0-2)).
Description: as for outcome 13
Time Frame: Baseline and Week 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg·hr/dL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 67 | 75 | 74
mg·hr/dL | -4.3 (60.23) | -74.7 (61.76) | -76.8 (63.19)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -70.38, 95% CI 2-sided [-90.67 to -50.09]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -72.49, 95% CI 2-sided [-93.10 to -51.88]

15. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing (AUC(0-2).
Description: The change between the value of insulin collected at week 12 or final visit and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 12
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: μU·hr/mL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 63 | 70 | 71
μU·hr/mL | -2.47 (10.817) | 4.62 (16.599) | 1.50 (14.845)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 7.093, 95% CI 2-sided [2.229 to 11.958]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 3.967, 95% CI 2-sided [-0.521 to 8.455]

16. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2).
Description: The change between the value of C-peptide collected at week 12 or final visit and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: ng·hr/mL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 68 | 75 | 74
ng·hr/mL | 0.14 (1.670) | 0.69 (1.901) | 0.57 (2.247)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.550, 95% CI 2-sided [-0.045 to 1.144]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = 0.428, 95% CI 2-sided [-0.233 to 1.090]

17. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)).
Description: The change between the value of glucagons collected at week 12 or final visit and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 12
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: pg·hr/mL
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 68 | 75 | 75
pg·hr/mL | -0.4 (64.18) | -19.2 (42.72) | -20.5 (41.97)
Statistical Analysis 1: Comparison: Voglibose 0.2 mg TID vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = -18.77, 95% CI 2-sided [-36.65 to -0.90]
Statistical Analysis 2: Comparison: Voglibose 0.2 mg TID vs Alogliptin 25 mg QD and Voglibose 0.2 mg TID; Test type: Superiority or Other; Mean Difference (Final Values) = -20.04, 95% CI 2-sided [-37.82 to -2.27]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Voglibose 0.2 mg TID | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Serious Adverse Events (participants affected / at risk) | 9/75 | 0/76 | 1/79
Other Adverse Events (participants affected / at risk) | 7/75 | 18/76 | 13/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voglibose 0.2 mg TID (N=75) | Alogliptin 12.5 mg QD (N=76) | Alogliptin 25 mg QD and Voglibose 0.2 mg TID (N=79)
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Blood and lymphatic system disorders) | 1 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voglibose 0.2 mg TID (N=75) | Alogliptin 12.5 mg QD (N=76) | Alogliptin 25 mg QD and Voglibose 0.2 mg TID (N=79)
Nasopharyngitis (Infections and infestations) | 4 | 17 | 13
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.